CLINICAL TRIAL: NCT06516874
Title: A Pilot Study of Feasibility and Acceptability of Videoconference-Delivered Trauma-Focused Cognitive Behavioral Therapy for Treatment of PTSD and C-PTSD in Adults of Community and Hospitals Mental Health Services
Brief Title: A Pilot Study of Trauma-Focused Cognitive-Behavioral Therapy for Treatment of Post-traumatic Stress in Adults.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Talca (Other)
Collaborators: Fondo Nacional de Desarrollo Científico y Tecnológico, Chile (Other Government); Universidad del Desarrollo (Other); Universidad Católica del Maule (Other); Servicio de Salud del Maule, Chile (Unknown)
Responsible Party: Principal Investigator, Andrés Fresno Rodríguez, Profesor Asociado, University of Talca
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FONDECYT REGULAR 1230715
Record Dates: First submitted 2024-07-02; First posted 2024-07-24 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Post Traumatic Stress Disorder; Complex Post-Traumatic Stress Disorder
Keywords: Pilot Study; Feasibility; Acceptability; Trauma-Focused Cognitive Behavioral Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: This study is a superiority pilot/feasibility study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trauma-Focused Cognitive Behavioral Therapy for complex presentation (TF-CBT-CP) (Experimental): The TF-CBT-CP includes: a) conducting clinical assessment sessions; b) providing psychoeducation on PTSD and CPTSD; c) facilitating the development of coping strategies to manage distressing experiences; d) implementing behavioral activation techniques to reintegrate into daily activities; e) fostering the acquisition of emotional regulation strategies and interpersonal relationship skills; f) utilizing in-vivo (live) and imaginal exposure methods to confront the traumatic memory; g) cognitive work to cope with distorted thoughts, and h) relapse prevention.
  Interventions: Behavioral: Trauma-Focused Cognitive Behavioral Therapy for complex presentation (TF-CBT-CP)

INTERVENTIONS:
Behavioral: Trauma-Focused Cognitive Behavioral Therapy for complex presentation (TF-CBT-CP) — This TF-CBT-CP is a short-term intervention to treat outpatients. This will be carried out via videoconference.

SUMMARY:
Post-traumatic stress disorder (PTSD) is a mental health condition that's triggered by the experience of potentially traumatic events. Complex PTSD (CPTSD) includes additional symptoms that account for a disturbance of the organization of the self. Randomized controlled trials have shown that trauma-focused cognitive behavioral therapy (TF-CBT) is effective in reducing PTSD symptoms; however, there is insufficient evidence to support the effectiveness of this intervention for CPTSD.

The present study aims to evaluate the feasibility and acceptability of TF-CBT therapy for complex presentation (TF-CBT-CP) in a videoconference modality in adults diagnosed with PTSD or CPTSD who are treated at community mental health care services (CMHCS, COSAM in Spanish) and the Hospital of the Maule Region, Chile.

This pilot study will use a mixed design. The quantitative component will consist of a one-group pre-post-follow-up design, which will include 13 adults diagnosed with PTSD or CPTSD referred to care at CMHCS or hospitals of the Maule Region, Chile. Telephone interviews will collect qualitative data relevant to the study's acceptability.

Participants will receive TF-CBT-CP therapy. It consists of 16 weekly 60-minute sessions of trauma-focused cognitive behavioral therapy for complex presentations.

To determine the feasibility of TF-CBT-CP therapy, eligibility, recruitment, participation, activity completion, retention, exit, and dropout rates will be considered. To establish the acceptability of the protocol, participant satisfaction with the recruitment, assessment, and treatment process and reporting of reasons for non-participation or dropout will be assessed. Furthermore, secondary outcomes consider the reduction of PTSD and CPTSD symptomatology, depression, and anxiety and the improvement of indicators of emotional regulation and psychological well-being.

DETAILED DESCRIPTION:
Post-traumatic stress disorder (PTSD) is a mental health condition that's triggered by the experience of potentially traumatic events. It is a disabling psychopathology with high comorbidity, associated with problems of emotional regulation and low psychological well-being. In addition, the World Health Organization (WHO) has recently proposed the diagnosis of complex PTSD (CPTSD) to account for a type of PTSD that includes both traditional and additional symptoms that account for a disturbance of self-organization of the self.

Randomized controlled trials (RCT) have shown that trauma-focused cognitive behavioral therapy (TF-CBT) is effective in reducing PTSD symptoms. However, additional clinical studies are necessary to fully assess the effectiveness of TF-CBT for complex presentations (TF-CBT-CP). Additionally, adapting PTSD therapy to a new population requires prior knowledge of information that may affect the effects of the intervention, e.g., history of traumatic events, variety and intensity of PTSD symptoms, and comorbidities. Given the lack of knowledge of these characteristics in Chile and for the purpose of subsequently implementing a large-scale randomized clinical trial in the Chilean population, the CONSORT guidelines recommend developing a pilot RCT.

The present study aims to evaluate the feasibility and acceptability of TF-CBT-CP therapy in a videoconference modality in adults diagnosed with PTSD or CPTSD who are treated at community mental health care services (CMHCS) or hospitals in the Maule Region, Chile. This pilot study will use a mixed design. The quantitative component will consist of a one-group pre-post-follow-up design, which will include 13 adults diagnosed with PTSD or CPTSD referred to care at CMHCS or hospitals of the Maule Region, Chile. Participants will receive-by videoconference-TF-CBT-CP therapy, which consists of 16 weekly 60-minute sessions of trauma-focused cognitive behavioral therapy for complex presentations.

The treatment includes a) conducting clinical assessment sessions; b) providing psychoeducation on PTSD and CPTSD; c) facilitating the development of coping strategies to manage distressing experiences; d) implementing behavioral activation techniques to reintegrate into daily activities; e) fostering the acquisition of emotional regulation strategies and interpersonal relationship skills; f) utilizing in-vivo (live) and imaginal exposure methods to confront the traumatic memory; g) engaging in cognitive interventions to address distorted thoughts; and h) implementing relapse prevention strategies. Clinical psychologists, trained by the research team, will implement the treatment. To ensure the fidelity of the TF-CBT-CP treatment, the project team will conduct weekly supervisions and review compliance with the activities of each session using a checklist based on the therapy protocol. The project team will provide supervision.

Professionals designated by CMHCS or hospitals will present the study to eligible individuals and ask if they are willing to be contacted by the study's research assistant(s) via telephone as part of the initial recruitment process. The research assistants will explain the study characteristics and the selection process, paying particular attention to the study inclusion and exclusion criteria. If the person agrees to participate, he or she will be invited to an in-person interview at the respective health services to address any doubts about the study and to complete the informed consent process.

Those who have agreed to participate and signed the informed consent form do the initial evaluation. This initial assessment will be conducted via videoconference, where trained psychologists will administer the Life Event Checklist-5 (LEC-5) and the International Trauma Questionnaire (ITQ), a self-report questionnaire that assesses PTSD and CPTSD symptoms. Trained psychologists administer the Mini-International Neuropsychiatric Interview (MINI) to determine whether individuals at risk for PTSD or CPTSD on previous instruments meet exclusion criteria. If the person is at risk of PTSD or CPTSD and does not meet any exclusion criteria, trained psychologists administer additional questionnaires to assess depressive (Patient Health Questionnaire, PHQ-9) and anxious symptoms (Generalized Anxiety Disorder Questionnaire, GAD-7), suicidal ideation and behavior (Columbia-Suicide Severity Rating Scale, C-SSRS), alcohol consumption and/or dependence (Alcohol and Other Drugs Use Questionnaire, AUDIT), emotional regulation problems (Spanish version of Difficulties in Emotion Regulation Scale, DERS-S), and impaired functioning (Work and Social Adjustment Scale, WSAS, and Clinical Outcomes in Routine Evaluation, CORE-10). In addition, another evaluation session is scheduled, where the diagnosis of PTSD or CPTSD is established through the International Trauma Interview (ITI). Participants who are excluded during this evaluation process will be invited to a feedback interview via videoconference.

Participants who meet the inclusion criteria and do not present exclusion criteria will engage in 16 weekly 60-minute sessions of trauma-focused cognitive behavioral therapy (TF-CBT-CP) through videoconference.

Participants will be invited to an evaluation session via video conference at the end of week 16 (final measurement) and week 20 (follow-up) after the start of treatment. During this session, they will participate in the International Trauma Interview (ITI) and complete the following questionnaires: ITQ, PHQ-9, GAD-7, C-SSRS, AUDIT, DERS-S, WSAS, and CORE-10. Furthermore, the participants' satisfaction with the intervention will be assessed using the Client Satisfaction Questionnaire (CSQ-8) at each of these measurement points.

To guarantee access to a computer with connectivity for video conferencing and a confidential space for TF-CBT-CP therapy, both the evaluation and treatment sessions will take place in the respective health services' room or in a similar clinical care center, where a notebook, internet connection, printer, camera, and microphone will be available to be used by study participants.

Trained psychologists will collect qualitative data related to the study's acceptability through telephone interviews after the follow-up measurement. They will apply an open-ended interview to all participants. Data collection will continue until the saturation point is reached. The thematic analysis will be done on the transcribed interviews.

To determine the feasibility of TF-CBT-CP therapy, eligibility, recruitment, participation, activity completion, retention, exit, and dropout rates will be considered. To establish the acceptability of the protocol, participant satisfaction with the recruitment, assessment, and treatment process and reporting of reasons for non-participation and dropout will be assessed. Secondary outcomes consider the reduction of PTSD and CPTSD symptomatology, depression, and anxiety, and the improvement of indicators of emotional regulation and psychological well-being.

ELIGIBILITY:
Eligibility criteria:

* Men and women over 18 years of age.
* Referred to a community mental health care service (CMHCS) or hospital in the Maule Region for difficulties associated with the experience of traumatic events, symptomatology, or diagnosis of Post-Traumatic Stress Disorder (PTSD) or the complex form of Post-Traumatic Stress Disorder (CPTSD).
* Not being treated for PTSD or C-PTSD at the time of recruitment

Inclusion Criteria:

* Men and women over 18 years of age.
* Referred to a community mental health care service (CMHCS) or hospital in the Maule Region for difficulties associated with the experience of traumatic events, symptomatology, or diagnosis of Post-Traumatic Stress Disorder (PTSD) or Complex Post-Traumatic Stress Disorder (CPTSD).
* Having the diagnosis of Post-Traumatic Stress Disorder (PTSD) or Complex Post-Traumatic Stress Disorder (CPTSD) by International Trauma Interview (ITI).
* Fluent in oral and written Spanish language.
* Access to telephone.

Exclusion Criteria:

* Previously or currently diagnosed psychotic disorder.
* Current substance use disorder.
* Current suicidal crisis.
* Depression is the primary diagnosis.
* Participation in a PTSD psychological treatment parallel to the study.

Study's exit criteria:

* Initiation of a psychological or pharmacological treatment for PTSD parallel to the study.
* Change of medication dose in the case of participants with pharmacological treatment prior to the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Eligibility rate as a feasibility indicator | At the baseline assessment during the recruitment period.
  Proportion of patients who meet eligibility criteria compared to the total number of patients registered in the community mental health care services and hospital referral system during the recruitment period.
Recruitment rate as a feasibility indicator. | At the baseline assessment during the recruitment period.
  The proportion of patients who accept the invitation to participate in the study with respect to those who meet the eligibility criteria.
Participation rate in the evaluation protocol as a feasibility indicator. | At baseline, 16-weeks and 20- week after the start of treatment.
  Proportion of patients who fully conclude activities in all 3 assessments: initial evaluation, at week 16 after the start of treatment (or end of treatment), and follow-up at week 20 after the start of treatment, with respect to the total number of people who agree to participate in the study.
Trauma-Focused Cognitive Behavioral Therapy for complex presentation (TF-CBT-CP) activities completion rate. | During the intervention period.
  Percentage of participants who concluded all (100%) of the proposed activities in the 16 treatment sessions, as reported in the TF-CBT-CP patients' activities diary carried out inside or outside sessions.
Participants retention rate as a feasibility indicator. | When the intervention is finished at 16 weeks after the start of treatment and at follow-up measurement (20 weeks after the start of treatment).
  Percentage of participants who remain in the study at weeks 16 and 20 after the start of treatment, respect to the total number of participants who started treatment.
Participants exit rate as a feasibility indicator. | When the intervention is finished at 16-weeks after the start of treatment and at follow-up measurement (20 weeks after the start of treatment).
  Proportion of participants who meet study exit criteria at weeks 16 and 20 after the start of treatment, compared to the total number of participants who started treatment.
Participants attrition rate as a feasibility indicator. | When the intervention is finished at 16 weeks after the start of treatment and at follow-up measurement (weeks after the start of treatment).
  Proportion of participants who drop out of the study at weeks 16 and 20 after the start of treatment, compared to the total number of participants who started treatment.
Qualitative description of the participants' acceptability as an acceptability indicator. | At follow-up measurement (20 weeks after the start of treatment).
  To obtain a qualitative description of participants' acceptability of the recruitment process, the assessment protocol (baseline, end-of-treatment, and follow-up assessment), and the treatment, semi-structured interviews will be conducted with participants, including questions related to acceptability of the study. The information collected will be recorded and summarized using thematic analysis guidelines.
Reasons for study refusals as an acceptability indicator | During the recruitment period.
  A list of reasons given by patients who refused to participate in the study. We will aggregate the results as percentages.
Reasons for study drop out as an acceptability indicator | During treatment (between week 1 and week 16 after starting treatment) and follow-up (20 weeks after starting treatment)
  A list of reasons given by patients who decided to drop-out the study. We will aggregate the results as percentages.
Participant satisfaction as an acceptability indicator | When the intervention is finished at 16 weeks after the start of treatment and at follow-up measurement (20 weeks after the start of treatment).
  Description of participant satisfaction level based on the Client Satisfaction Questionnaire (CSQ-8). The CSQ-8 is a self-report scale of 8 items that evaluate patients' overall satisfaction with treatment through a Likert scale from 1 (low satisfaction) to 4 (high satisfaction); the higher the score, the higher the patients' satisfaction.

SECONDARY OUTCOMES:
Changes in PTSD symptoms, according to mean scores obtained with the International Trauma Questionnaire (ITQ). | At baseline, 16 weeks, and 20 weeks after the start of treatment.
  The ITQ (International Trauma Questionnaire) is an 18-item self-report scale that assesses PTSD and complex PTSD (CPTSD) symptomatology based on the International Classification of Diseases 11 (ICD-11) and functional impairment. Each item is scored on a Likert scale ranging from 0 (not at all) to 4 points (extremely); the higher the score, the greater the symptomatology.
Changes in CPTSD symptoms, according to mean scores obtained with the International Trauma Questionnaire (ITQ). | At baseline, 16 weeks, and 20 weeks after the start of treatment.
  The ITQ (International Trauma Questionnaire) is an 18-item self-report scale that assesses PTSD and complex PTSD (CPTSD) symptomatology based on the International Classification of Diseases 11 (ICD-11) and functional impairment. Each item is scored on a Likert scale ranging from 0 (not at all) to 4 points (extremely); the higher the score, the greater the symptomatology.
Changes in PTSD symptoms, according to mean scores obtained with the International Trauma Interview (ITI). | At baseline, 16 weeks, and 20 weeks after the start of treatment.
  The ITI (International Trauma Interview) is a 16-item semi-structured interview that allows for determining the diagnosis of PTSD and CPTSD by assessing PTSD symptoms and Disturbances in Self-Organization symptoms. The interview takes between 45 and 60 minutes.
Changes in CPTSD symptoms, according to mean scores obtained with the International Trauma Interview (ITI). | At baseline, 16 weeks, and 20 weeks after the start of treatment.
  The ITI (International Trauma Interview) is a 16-item semi-structured interview that allows for determining the diagnosis of PTSD and CPTSD by assessing PTSD symptoms and Disturbances in Self-Organization symptoms. The interview takes between 45 and 60 minutes.
Change in depressive symptoms according to mean scores obtained with the Patient Health Questionnaire (PHQ-9). | At baseline, 16 weeks, and 20 weeks after the start of treatment.
  The PHQ-9 is a 9-item self-report scale assessing the frequency of depressive symptoms in the past 2 weeks. Its response scale is 0 = "never," 1 = "some days," 2 = "more than half of the days," and 3 = "almost every day." The higher the score, the greater the symptomatology. This scale has been translated and validated for the Chilean population.
Change in anxiety symptoms according to mean scores obtained with the Generalized Anxiety Disorder Questionnaire (GAD-7). | At baseline, 16 weeks, and 20 weeks after the start of treatment.
  The GAD-7 is a 7-item self-report scale assessing the frequency of anxious symptoms during the past 2 weeks. Its response scale is 0 = "not at all," 1 = "several days," 2 = "more than half of the days," and 3 = "nearly every day." The higher the score, the greater the symptomatology.
Change in emotion regulation according to mean scores obtained with the Spanish version of the Difficulties in Emotion Regulation Scale (DERS-S). | At baseline, 16 weeks, and 20 weeks after the start of treatment.
  The DERS-S is a 25-item self-report scale that assesses emotional regulation problems. Its Likert-type response scale ranges from 1 (almost never) to 5 (almost always). The lower the score, the better emotion regulation.
Change in psychological well-being as measured by the Work and Social Adjustment Scale ("WSAS") score. | At baseline, 16 weeks, and 20 weeks after the start of treatment.
  The WSAS is a 5-item self-report scale that assesses impairment in functioning, considering the impact of a person's mental health difficulties on their ability to function in terms of work, home management, social leisure, private leisure, and personal or family relationships. The higher the score, the greater the functional impairment.
Change in psychological well-being as measured by the Clinical Outcomes in Routine Evaluation (CORE-10) score. | At baseline, 16 weeks, and 20 weeks after the start of treatment.
  The CORE-10 is a self-reported 10-item measure for common presentations of psychological distress. The higher the score, the higher the psychological distress.
Change in psychological well-being as measured by the International Trauma Questionnaire (ITQ) impairment items. | At baseline, 16 weeks, and 20 weeks after the start of treatment.
  International Trauma Questionnaire (ITQ) items associated with impairment in important areas of functioning refer to items that assess impairment in the person's functioning associated with PTSD symptoms or DSO symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Andrés Fresno Rodríguez, Principal Investigator — University of Talca
Locations (5):
- Chile (5):
  - Centro Comunitario de Salud Mental de Curicó (COSAM), Curicó, Maule Region
  - Centro Comunitario de Salud Mental de Linares (COSAM), Linares, Maule Region
  - Hospital de Linares, Linares, Maule Region
  - Centro Comunitario de Salud Mental de Maule (COSAM), Maule, Maule Region
  - Centro Comunitario de Salud Mental de Talca (COSAM), Talca, Maule Region

IPD SHARING:
Plan to Share IPD: No
The approval by the ethics committee did not contemplate the possibility of sharing individual patient data (IPD)